CLINICAL TRIAL: NCT06888765
Title: The Impact of Changes in Body Composition on the Retina and Choroid
Brief Title: Effects of Differences in Body Composition on Retina and Choroid
Status: Completed | Type: Observational
Sponsor: Bayram Meydan (Other)
Responsible Party: Sponsor-Investigator, Bayram Meydan, Research Assistant, MD, Duzce University
Organization: Duzce University (Other)
Other Study IDs: ETHICS-2024-113; 2024-113 (Other: Düzce University Non-Interventional Ethics Committee)
Record Dates: First submitted 2025-03-07; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Obesity, Morbid; Body Composition
Keywords: Obesity; Retina; Choroid; Body Mass Index (BMI); Body Composition Analysis; Optical Coherence Tomography (OCT); Microvascular Structures
MeSH Terms: conditions — Obesity; Obesity, Morbid | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Underweight: Participants with BMI <18.5
  Interventions: Other: Optical Coherence Tomography (OCT) and Body Composition Analysis
- Normal Weight: Participants with BMI between 18.5 and 24.9
  Interventions: Other: Optical Coherence Tomography (OCT) and Body Composition Analysis
- Overweight: Participants with BMI between 25 and 29.9
  Interventions: Other: Optical Coherence Tomography (OCT) and Body Composition Analysis
- Obese: Participants with BMI between 30 and 34.9
  Interventions: Other: Optical Coherence Tomography (OCT) and Body Composition Analysis
- Severely Obese: Participants with BMI >35
  Interventions: Other: Optical Coherence Tomography (OCT) and Body Composition Analysis

INTERVENTIONS:
Other: Optical Coherence Tomography (OCT) and Body Composition Analysis — This observational study included non-invasive diagnostic assessments to evaluate retinal, choroidal, ocular, and body composition parameters. Optical Coherence Tomography (OCT) measured macular and peripapillary retinal parameters, including retinal volume and cup/disc ratio. Enhanced Depth Imaging OCT (EDI-OCT) assessed choroidal thickness and vascularity, while Optical Coherence Tomography Angiography (OCTA) analyzed vessel density and foveal avascular zone (FAZ) metrics.
  Optical biometry measured axial length, anterior chamber depth, lens thickness, K1, K2, and central corneal thickness. Autorefractometry and tonometry were part of the routine ophthalmologic examination, including slit-lamp biomicroscopy. Bioelectrical impedance analysis (BIA) assessed body composition, including BMI, fat percentage, muscle mass, and metabolic age. These assessments were for research purposes only, without therapeutic intervention.

SUMMARY:
The goal of this observational study is to examine the effects of body composition differences on retinal and choroidal structures. The study aims to investigate how variations in fat distribution and body composition parameters influence ocular microvascular structures.

The main questions it aims to answer are:

* How do differences in body composition (BMI, waist circumference, bioelectrical impedance parameters) affect retinal and choroidal microvascular structures?
* Are there significant structural changes in the retina and choroid among individuals with different body composition profiles?

Participants will:

* Be classified into five groups based on their Body Mass Index (BMI) (underweight, normal weight, overweight, obese, and severely/morbidly obese).
* Undergo detailed body composition analysis using bioelectrical impedance analysis (BIA) to assess fat mass, muscle mass, visceral fat index, and metabolic age.
* Receive comprehensive ophthalmologic evaluations, including Optical Coherence Tomography (OCT) and Optical Coherence Tomography Angiography (OCTA), to measure retinal thickness, choroidal thickness, and microvascular parameters.
* OCTA images will be analyzed using the OCTAVA software to compute vascular parameters.

This study does not involve any new treatments, drugs, or interventional procedures. The findings aim to provide insights into the relationship between body composition and ocular microvascular health, contributing to early detection and prevention strategies for obesity-related ocular complications.

DETAILED DESCRIPTION:
Study Overview

This study is a prospective observational research planned to be conducted at Düzce University between July 1, 2024, and October 1, 2024. The aim of this study is to evaluate the potential effects of body composition differences on retinal and choroidal microvascular structures using non-invasive imaging techniques. The study is designed to investigate how obesity-related changes in fat distribution, metabolic parameters, and vascular structures may influence ocular health.

A total of 200 participants are planned to be enrolled, consisting of individuals who will visit the ophthalmology clinic for routine eye examinations and will be confirmed to have no pre-existing ocular pathologies. Participants will be classified into five groups based on Body Mass Index (BMI):

* Group 1: Underweight (BMI <18.5)
* Group 2: Normal weight (BMI 18.5-24.9)
* Group 3: Overweight (BMI 25-29.9)
* Group 4: Obese (BMI 30-34.9)
* Group 5: Severely/Morbidly Obese (BMI >35)

Each group is expected to include 40 participants.

Planned Study Procedures and Measurements Ophthalmologic Evaluations

All participants will undergo a comprehensive ophthalmologic examination, including:

* Autorefractometry to assess refractive errors
* Intraocular pressure (IOP) measurement using a non-contact tonometer
* Detailed slit-lamp biomicroscopy to examine anterior and posterior segment structures Body Composition Analysis
* Bioelectrical Impedance Analysis (BIA) will be performed to assess:
* Total body fat percentage, visceral fat index, muscle mass, and metabolic age
* Segmental body composition (fat and muscle mass in arms, legs, and trunk)
* Extracellular and intracellular water distribution
* Waist circumference, waist-to-hip ratio, waist-to-height ratio OCT and OCTA Imaging
* Optical Coherence Tomography (OCT) and Enhanced Depth Imaging-OCT (EDI-OCT) will be used to obtain:
* Macular and peripapillary retinal thickness measurements
* Retinal nerve fiber layer (RNFL) thickness
* Optic disc and cup-to-disc ratio analysis
* Choroidal thickness at the subfoveal region and 500 µm intervals
* Optical Coherence Tomography Angiography (OCTA) will be performed to analyze:
* Superficial and deep retinal capillary plexus vascular density
* Foveal avascular zone (FAZ) area, perimeter, and circularity
* Vascular tortuosity and branchpoint density Image Processing and Analysis
* OCTA images will be analyzed using the OCTAVA software, where:
* Vessel area density, vessel length density, total vessel length, mean vessel diameter, median vessel diameter, branchpoint density, fractal dimension, and vessel tortuosity will be calculated.
* FAZ metrics (FAZ area, perimeter, and circularity) and vascular density values will be evaluated using ETDRS grid segmentation and FD-300 analysis.
* Choroidal Vascularity Index (CVI) will be calculated from EDI-OCT images using ImageJ software.

Study Objectives and Clinical Significance

This study aims to determine the relationship between body composition differences and retinal/choroidal microvascular changes to better understand how systemic metabolic alterations influence ocular structures. The results are expected to contribute to:

* Identifying early ocular biomarkers associated with obesity
* Developing preventive strategies for obesity-related retinal and choroidal complications
* Enhancing the clinical use of non-invasive imaging techniques in metabolic disease monitoring No new treatment, drug, or interventional procedure is planned to be applied in this study, and no life-threatening risks are anticipated.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years,
* No detected pathology in routine ophthalmologic examination,
* Providing written informed consent for participation.

Exclusion Criteria:

* Presence of ocular diseases such as glaucoma, uveitis, diabetic retinopathy, amblyopia, or retinal vein occlusion,
* History of previous ocular surgery,
* Refractive error exceeding ±4 diopters,
* Use of medications that may affect choroidal or retinal vascular structures,
* Pregnancy or breastfeeding,
* Presence of metallic prostheses, pacemakers, or other implants that could interfere with body composition analysis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study aims to evaluate changes in ocular microvascular structures in healthy individuals aged 18-65 years with different body mass index (BMI) categories. Participants included in the study have no systemic or ophthalmologic diseases, and their refractive error is within the ±4 diopter range.
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Central Macular Thickness (CMT) | Baseline (Cross-sectional)
  Measurement of central macular thickness (CMT) in micrometers using spectral-domain Optical Coherence Tomography (OCT). The measurement focuses on the 1 mm central foveal region.
Peripapillary Retinal Nerve Fiber Layer (RNFL) Thickness | Baseline (Cross-sectional)
  Measurement of peripapillary RNFL thickness in micrometers using spectral-domain OCT. RNFL thickness is assessed around the optic disc at baseline.
Choroidal Thickness | Baseline (Cross-sectional)
  Subfoveal choroidal thickness (in micrometers) measured using Enhanced Depth Imaging OCT (EDI-OCT). Measurements are taken at the fovea and at predefined intervals (e.g., 500 µm, 1000 µm) on either side of the fovea.
Choroidal Vascularity Index (CVI) | Baseline (Cross-sectional)
  Calculation of the choroidal vascularity index (CVI) as the ratio of luminal area to total choroidal area in EDI-OCT images. Measurements are performed at the subfoveal region and analyzed using ImageJ software.
Retinal Microvascular Parameters (OCTA) | Baseline (Cross-sectional)
  Evaluation of retinal microvascular parameters using Optical Coherence Tomography Angiography (OCTA). Metrics include vascular density, vessel length, and foveal avascular zone (FAZ) area/circularity in both superficial and deep capillary plexuses.

SECONDARY OUTCOMES:
Composite Association Between Body Composition and Ocular Parameters | Baseline
  This composite outcome measure includes correlation analyses between BIA parameters (fat percentage, muscle mass, visceral fat, metabolic rate) and multiple ocular structures (central macular thickness, RNFL thickness, choroidal thickness, CVI). The aim is to determine whether body composition influences overall microvascular integrity.
Composite Regional Vascular Density Changes in Retinal and Choroidal Layers | Baseline
  This composite outcome measure evaluates retinal and choroidal vascular densities (VAD, VLD) in predefined ETDRS regions (foveal, parafoveal, perifoveal) using OCTA. The objective is to compare these densities across different BMI groups.

OTHER OUTCOMES:
FAZ Area | Baseline
  Measurement of the foveal avascular zone (FAZ) area (in mm²) using OCT Angiography to evaluate differences across BMI groups.
FAZ Perimeter | Baseline
  Measurement of the FAZ perimeter (in mm) using OCT Angiography to assess potential variations in foveal microcirculation among different BMI categories.
FAZ Circularity Index | Baseline
  Assessment of FAZ shape using a circularity index. Higher values indicate a more circular FAZ. Comparisons will be made across underweight, normal, overweight, obese, and severely obese groups.
Axial Length | Baseline
  Comparison of axial length measurements among different BMI categories to identify possible associations with ocular morphology.
Autorefraction Measurements | Baseline
  Spherical equivalent refraction (in diopters) measured using an autorefractometer. Differences across BMI categories will be assessed.
Intraocular Pressure Measurements | Baseline
  Intraocular pressure (IOP) measured in mmHg using a non-contact tonometer. Differences across BMI groups will be evaluated.
Anthropometric Measurements (Waist, Hip, and Height) | Baseline
  This outcome measure includes the measurement of waist circumference, hip circumference, and height. From these, waist-to-hip ratio (WHR) and waist-to-height ratio (WHtR) are calculated to assess central obesity. All measurements are performed following standardized protocols at baseline.
Body Composition Analysis | Baseline
  This outcome measure involves the analysis of body composition parameters using bioelectrical impedance analysis (BIA) with the Tanita BC-418 MA device. Parameters such as body weight, body mass index (BMI), total fat percentage, muscle mass, visceral fat, and basal metabolic rate are recorded. These data are compared across different BMI groups to evaluate overall body composition differences.

CONTACTS AND LOCATIONS:
Overall Officials: MURAT KAYA, Prof. Dr., Principal Investigator — Duzce University Faculty of Medicine, Department of Ophthalmology; BAYRAM MEYDAN, MD, Research Assistant, Principal Investigator — Duzce University Faculty of Medicine, Department of Ophthalmology
Locations (1):
- Duzce Univ. Fac. of Medicine, Dept. of Ophthalmology, Düzce, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical considerations and data privacy regulations. The collected data contain sensitive personal health information, and sharing them could potentially violate patient confidentiality and institutional policies. Additionally, there are no plans for a public data repository for this study.

REFERENCES:
- [Background] Tapp RJ, Owen CG, Barman SA, Welikala RA, Foster PJ, Whincup PH, Strachan DP, Rudnicka AR; UK Biobank Eye, Vision Consortium. Retinal Vascular Tortuosity and Diameter Associations with Adiposity and Components of Body Composition. Obesity (Silver Spring). 2020 Sep;28(9):1750-1760. doi: 10.1002/oby.22885. Epub 2020 Jul 29. PMID 32725961
- [Background] Ozgur G, Gokmen O. Associations between body mass index and choroidal thickness, superficial and deep retinal vascular indices, and foveal avascular zone measured by OCTA. Photodiagnosis Photodyn Ther. 2023 Jun;42:103515. doi: 10.1016/j.pdpdt.2023.103515. Epub 2023 Mar 14. PMID 36924979
- [Background] Dogan B, Dogan U, Gedik B, Turkmen B, Cakir RC, Demirer ME, Aslaner A. Optical coherence tomography angiography evaluation of optic disc and retinal vascular densities in obese patients. Photodiagnosis Photodyn Ther. 2023 Dec;44:103826. doi: 10.1016/j.pdpdt.2023.103826. Epub 2023 Oct 4. PMID 37797912